CLINICAL TRIAL: NCT03411967
Title: Clinical Study of Apatinib in Combination With Docetaxel for Patients With Advanced NSCLC After Failure of Platinum-based Double-drug Therapy
Brief Title: Apatinib in Combination With Docetaxel for Patients With Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zigong No.1 Peoples Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APTN-L201712
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — apatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib combine with docetaxel (Experimental): Docetaxel, 60 mg / m2, d1, iv + apatinib 500mg, po, qd
  Interventions: Drug: Apatinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Apatinib — apatinib mesylate tablets 500mg, po, qd, continued until the next cycle, taking on an empty stomach (daily taken at the same time), every 3 weeks For one cycle, a total of 4 to 6 cycles of treatment, apatinib has been taken until the disease progresses, intolerable toxicity.
  Other Names: Aitan
Drug: Docetaxel — Docetaxel, 60 mg / m2, d1, iv ,every 3 weeks For one cycle, a total of 4 to 6 cycles of treatment

SUMMARY:
In order to explore a new treatment strategy for patients with failed NSCLC platinum-containing double-drug therapy, this study was to investigate the clinical efficacy of apatinib in combination with docetaxel for patients with advanced NSCLC after failure of platinum-based regime

ELIGIBILITY:
Inclusion Criteria:

1. ECOG 0-2;
2. Expected survival of not less than 12 weeks;
3. The first line of platinum-containing chemotherapy, pathologically confirmed IIIB, IV non-small cell lung cancer, with measurable lesions (according to the RECIST 1.1 standard, CT lesion tumor diameter ≥ 10mm, lymph node lesion CT scan diameter ≥ 15mm, measurable lesions have not received radiotherapy, local treatment such as freezing)
4. The main organs function properly
5. Women of childbearing age must have had reliable contraception or have had a pregnancy test (serum or urine) within 7 days prior to enrollment with a negative result and are willing to take appropriate measures 8 weeks after and during the last administration of the test drug contraception. In the case of males, consent is to be given to contraception or surgical sterilization 8 weeks after and during the last administration of the test drug;
6. Participants volunteered to join the study and signed informed consent form, with good compliance and follow-up.

Exclusion Criteria:

1. Imaging (CT or MRI) showed tumor lesions away from the large blood vessels ≤ 5mm, or the presence of invasive central local blood vessels of the central tumor; or showed the presence of significant lung empty or necrotic tumors;
2. Uncontrolled hypertension (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg, despite optimal drug therapy);
3. Has the following cardiovascular disease: Myocardial ischemia or myocardial infarction with grade II or higher, poorly controlled arrhythmia (including QTc intercourse men ≥ 450ms, women ≥ 470ms); NYHA class III-IV cardiomyopathy, Or cardiac ultrasound examination prompted left ventricular ejection fraction (LVEF) <50%;
4. Hemoptysis (INR> 1.5 or Prothrombin Time (PT)> ULN + 4 seconds or APTT> 1.5ULN) with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
5. In the first 2 months before enrollment, there is obvious slightly blood, or daily hemoptysis volume of 2.5ml or more;
6. Within 3 months prior to enrollment, significant clinically significant bleeding symptoms or definite bleeding tendencies such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ at baseline, and above, or vasculitis;
7. Incidence of arterial / venous thrombosis within the first 12 months of enrollment such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
8. Known hereditary or acquired bleeding and thrombophilia (eg hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc);
9. Factors that significantly affect the absorption of oral drugs, such as non-swallowing, chronic diarrhea and intestinal obstruction;
10. Urine routine urinary protein ≥ ++, or confirmed 24-hour urinary protein content ≥ 2.0g;
11. Previous or concurrent with other unhealed malignancies, except for those having had a cure for cutaneous basal cell carcinoma, carcinoma of the cervix, and superficial bladder cancer;
12. Pregnant or lactating women; Reproductive patients who are unwilling or unable to take effective contraception;
13. The investigators determine other situations that may affect clinical research and outcome decisions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 month
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | 12 month
  Progress-Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: 132100694 132100694, M.D., Principal Investigator — Zigong No.1 People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided